CLINICAL TRIAL: NCT02632084
Title: Follow-up Evaluation of Photo-Dynamic Therapy for Pituitary Tumours
Status: Completed | Type: Observational
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: NE13/10696
Record Dates: First submitted 2015-12-10; First posted 2015-12-16 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Pituitary Neoplasms
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
A study to followup patients that have previously been treated for pituitary tumours with either photodynamic therapy or placebo in a previous trial. The study aims to determine whether photodynamic therapy has any long term effect on tumour size, visual fields or endocrinological function.

DETAILED DESCRIPTION:
No patients will receive any medical or procedural treatments in this study, since these have been administered in a previous trial. The previous trial participants will be contacted and asked to attend a clinic or to have a telephone interview, where they will answer a questionnaire. They will be assessed clinically for visual fields, as well as undergoing an MRI scan of their head to assess tumour size (unless they have had a scan anyway in the previous 12 months), these tests would ordinarily form part of the routine outpatient workup for patients with pituitary tumours. There is no significant risk to the physical well-being of the patients with any of the methods to be used.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were previously included in the initial pituitary PDT trial, in addition to those who were randomised as part of the RCT arm of the study. These patients have already participated in phase I/II trials. Of note, these patients all have pituitary tumours.

Exclusion Criteria:

* Patients who were not included in the above mentioned trials. Patients included in the original trials who have subsequently died (of any cause).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Details of previous research participants will be extracted from the study files by the researchers, who are all members of the direct care team.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Tumour size on MRI scan. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom